CLINICAL TRIAL: NCT03018327
Title: Ano-genital Human Papillomavirus (HPV) Infection, Genital Warts, Precancerous Lesions and Cancer Among Danish Renal Transplant Recipients
Brief Title: Ano-genital Human Papillomavirus (HPV) Infection, Precancerous Lesions and Genital Warts Among Danish Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Helle Kiellberg Larsen, Staff specialist, Bispebjerg Hospital
Other Study IDs: H-15014510
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Anogenital Dysplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — HPV samples tested by Inno-lipa
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case group: 250 Renal Transplant Recipients; 125 women and 125 men
- Control group: 250 healthy controls; 125 women and 125 men

SUMMARY:
Transplant-related malignancies have emerged as one of the important complications after organ transplantation. Some studies have shown that transplant recipients have an increased risk of developing cancer, especially non-melanoma skin cancer. Because of iatrogenic immunosuppression in these patients, there is an increasing focus on human papillomavirus (HPV) related cancers.

The occurrence of HPV infection and ano-genital precancerous lesions and genital warts among Danish renal transplant recipients (RTRs) is not known. Relatively few controlled studies exist on the prevalence of ano-genital HPV infection, anal precancerous lesions and cervical precancerous lesions among RTRs.

Knowledge about HPV infection and HPV-related ano-genital precancerous lesions in renal transplant recipients, together with identification of factors that play a role for development of anal and cervical precancerous lesions, is important for the possibility of early detection and treatment to prevent progression to ano-genital cancers. Cervical cytology has been used for decades to detect cervical intra-epithelial neoplasia (CIN), whereas high-resolution anoscopy is a newer modality for the detection of anal intra-epithelial neoplasia (AIN). International guidelines recommend annually screening against cervical cancer for female renal transplant recipients, but currently no recommendation exists on screening against anal cancer.

Aim: In a clinical study it is the aim to examine the prevalence of anal, penile, oral and cervical HPV infection as well as ano-genital dysplasia and ano-genital warts among 250 renal transplant recipients and an immunocompetent control group. Furthermore to identify factors associated with the development of AIN or CIN such as HPV type, viral load, duration of immunosuppression, and lifestyle factors such as sexual habits, reproductive history, smoking and alcohol habits, history of genital warts and other infections, and socio-economic variables.

ELIGIBILITY:
Inclusion Criteria:

-

Case group:

1. Renal transplant recipients men and women ≥ 18 years of age
2. ≥ 6 months posttransplantation
3. Stabile immunosuppressive regime
4. No signs of acute rejection og the transplant

Control group:

1. Health men and women ≥18years of age from the Nevus clinic, Laser clinic and non-melanoma skin cancer clinic, Bispebjerg Hospital, Copenhagen

Exclusion Criteria:

* Case group:

  1. Other known immunosuppression

     Both case- og control group:
  2. Previous HPV vaccination
  3. Previous total hysterectomy
  4. Inflammatory bowel disease
  5. HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will include 250 male and female renal transplant recipients in the case group. The patients will be recruited from "The Transplantation Clinic" at the Department of Dermato-venereology, Bispebjerg Hospital (BBH), where they are being followed for development of cutaneous (pre-)malignancies and from the Department of Nephrology at Rigshospital and Herlev Hospital, Denmark. In the control group we will include 250 immunocompetent individuals consisting of male and female patients coming for control of birthmarks at the Nevus Clinic or Non-melanoma skin cancer and precancer at BBH and patients having laser treatment for benign cutaneous lesions at BBH. The participants will be enrolled in the study after informed consent has been obtained.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-01-07; Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of ano-genital HPV infection, dysplasia and warts | 18 month
  Prevalence of oral, penile, cervical and anal HPV infection, ano-genital dysplasia and warts

SECONDARY OUTCOMES:
Risk factors for the development of ano-genital dysplasia and warts | 18 month
  Identifying factors associated with the development of AIN or CIN such as HPV type, viral load, duration of immunosuppression, and lifestyle factors such as sexual habits, reproductive history, smoking and alcohol habits, history of genital warts and other infections, and socio-economic variables.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Kiellberg Larsen, MD, Principal Investigator — Department of Dermato-venereology, Bispebjerg Hospital, 2400 Copenhagen, Denmark
Locations (1):
- Department of Dermato-venereology, Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Larsen HK, Kjaer SK, Haedersdal M, Kjaer AK, Bonde JH, Sorensen SS, Thomsen LT. Anal Human Papillomavirus Infection in Kidney Transplant Recipients Compared With Immunocompetent Controls. Clin Infect Dis. 2022 Nov 30;75(11):1993-1999. doi: 10.1093/cid/ciac285. PMID 35438132